CLINICAL TRIAL: NCT02577393
Title: Study of Epigallocatechin-3-gallate (EGCG) for Esophagus Protection in Patients With Lung Cancer Receiving Radial Radiotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Han Xi Zhao, Principal Investigator, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GTEEC-2015
Record Dates: First submitted 2015-09-28; First posted 2015-10-16 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Lung Neoplasms; Esophagitis; Prevention & Control; Epigallocatechin Gallate
Keywords: Lung Neoplasms; esophagitis; Prevention & Control; Epigallocatechin Gallate
MeSH Terms: conditions — Lung Neoplasms; Esophagitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- prophylactic EGCG group (Experimental)
  Interventions: Drug: EGCG
- therapeutic EGCG group (Experimental)
  Interventions: Drug: EGCG
- conventional therapy group (Placebo Comparator)
  Interventions: Drug: mLDG

INTERVENTIONS:
Drug: EGCG — EGCG (purity≥95% by high pressure liquid chromatography; from Ningbo HEP Biotech Co., Ltd) is dissolved in 0.9% saline solution three times a day. A new batch is made up each time. For esophageal application, repeated swallowing of 10 ml of the EGCG solution is indispensable to assure the prolonged presence of drug the esophageal walls. We choose a dose of 440 lmol/L as the recommended concentration for this study by referring to our previous phase I study. Immediately at the beginning of radiotherapy, the EGCG solution is given until two weeks after radiotherapy completed. Steroids, non-steroidal anti-inflammatory drugs, narcotics, local anesthetics, or other antibiotic/antifungal therapy are not given unless esophagitis progressed to grade 4.
  Arms: prophylactic EGCG group
Drug: EGCG — EGCG (purity≥95% by high pressure liquid chromatography; from Ningbo HEP Biotech Co., Ltd) is dissolved in 0.9% saline solution three times a day. A new batch is made up each time. For esophageal application, repeated swallowing of 10 ml of the EGCG solution is indispensable to assure the prolonged presence of drug the esophageal walls. We choose a dose of 440 lmol/L as the recommended concentration for this study by referring to our previous phase I study. Patients begin medications as soon as grade 1 esophagitis occurred during radiation according to the RTOG criterion.
  Arms: therapeutic EGCG group
Drug: mLDG — mLDG (lidocaine 0.16mg/mL, dexamethasone 0.02mg/mL, and gentamycin 0.16mg/mL) dissolved in 0.9% saline solution was administered three times a day. Patients were given oral mLDG solution, and began medications as soon as grade 1 esophagitis occurred during radiation according to the RTOG criterion.
  Arms: conventional therapy group

SUMMARY:
The investigators conducted this phase II study of EGCG therapy protection of the esophagus from damage induced by radiotherapy. In order to observe the effectiveness of EGCG, esophageal toxicity was recorded weekly using a grading scale based on symptomatology, following the Radiation Therapy Oncology Group (RTOG) scoring system. Patient-reported pain related to esophagitis was measured using the numerical rating scale (NRS) every week from EGCG application to 2 weeks after the end of radiotherapy. The scales are translated into Chinese and guides in Chinese are developed instructing how to use the scales and perform the assessments.

ELIGIBILITY:
Inclusion Criteria:

* pathologically documented LC
* considered medically inoperable stage IIIA or stage IIIB or limited stage small cell lung cancer
* age ≥18 years
* Karnofsky ≥70
* adequate hematologic, hepatic and renal function
* FEV1 > 800 cc
* mean esophagus dose >20 Gy

Exclusion criteria were as follows:

* a known allergy or hypersensitivity to EGCG
* pregnancy or lactation
* prior radiation to the thorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Superiority of EGCG in reducing Grade II esophagitis as assessed by RTOG scores in patients with lung cancer receiving radiation | Each patient will be enrolled for a 8-9 week trial

SECONDARY OUTCOMES:
Superiority of EGCG in decreasing the serum Inflammatory factors in patients with lung cancer receiving radiation | Each patient will be enrolled for a 8-9 week trial
Improved quality of life with usage of EGCG for treatment of radiation-esophagitis in patient with lung cancer. | Each patient will be enrolled for a 8-9 week trial

CONTACTS AND LOCATIONS:
Overall Officials: Ligang Xing, MD,PhD, Study Chair — Shandong Cancer Hospital and Institute